CLINICAL TRIAL: NCT01871077
Title: Phase I Clinical Trial to Assess the Safety and Tolerability of the Ophthalmic Solution PRO-156 Over the Ocular Surface of Ophthalmologically Healthy Volunteers.
Brief Title: Safety and Tolerability of the Ophthalmic Solution PRO-156 in Ophthalmologically Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOPH156-0612/I
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Results first posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Healthy
MeSH Terms: interventions — Ketorolac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRO-156 (Experimental): Drug: PRO-156 ophthalmic solution One drop of PRO-156 ophthalmic solution administered to each eye, four times a day for 10 days.
  Interventions: Drug: PRO-156

INTERVENTIONS:
Drug: PRO-156 — Drug: PRO-156 ophthalmic solution One drop of PRO-156 ophthalmic solution administered to each eye, four times a day for 10 days.
  Other Names: Ketorolac

SUMMARY:
The purpose of this study is to evaluate safety and tolerability of the ophthalmic solution PRO-156 over the ocular surface of ophthalmologically healthy volunteers

DETAILED DESCRIPTION:
A phase I, open label and unicentric clinical trial to evaluate the safety and tolerability of the ophthalmic solution PRO-143 over the ocular surface of ophthalmologically healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female.
* Age between 18 and 40 years old at screening visit.
* Signed informed consent

Exclusion Criteria:

* Patient with one blind eye.
* Any ocular or systemic condition.
* Visual acuity of 20/100 in any eye.
* Use of ocular or systemic medication.
* Contraindications or sensitivity to any component of the study treatment.
* Contact lens users.
* Ocular surgery within the past 3 months..
* Pregnant, nursing or childbearing potential women who were not using effective contraception.
* Participation in any studies of investigational drugs within 90 days previous to the inclusion.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Casillas, MD, Principal Investigator — Independent Clinical Research Center

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 32 ophthalmologically healthy volunteers were evaluated, to which both eyes, with no history of any systemic or ophthalmological disease, who were not using any type of medication, and who agreed to participate in the study and met all the inclusion criteria described in the section.
Pre-assignment Details: Only 30 were selected and 2 discarded because they met the exclusion criteria.
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | PRO-156
Started | 30; 60 eyes
Completed | 30; 60 eyes
Not Completed | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: The study population consisted of ophthalmologically healthy volunteers, with no history of any systemic or ophthalmological disease, with both ayes, who were not using any type of medication, and who agreed to participate in the study and met all the inclusion criteria described in the section and with none of the exclusion criteria.
Units Other Than Participants: eyes
Arm/Group | PRO-156
Number analyzed (Participants) | 30
Number analyzed (eyes) | 60
Age, Continuous [Median (Full Range); unit: years] | 27 [18 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0
  Race: Asian | 0
  Race: Native Hawaiian or Other Pacific Islander | 0
  Race: Black or African American | 0
  Race: White | 0
  Race: More than one race | 30
  Race: Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 30

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity (VA)
Description: The VA will be evaluated basally, without refractive correction with the Snellen chart. A Snellen chart is placed at a standard distance: 20 ft. At this distance, the symbols on the line representing "normal" acuity subtend. This line, designated 20/20 is the smallest line that a person with normal acuity can read at a distance of 20fs. the scale consists of 11 lines of letters of different size, the size of the letter gives a fractional value according to the visual acuity of the patient, the value is inversely proportional to the visual acuity, if the denominator is greater the visual acuity will be less.
  Line 1: 20/200 Line 2: 20/100, Line 3: 20/70, line 4: 20/50, line 5: 20/40, Line 6: 20/30, line 7: 20/25, Line 8: 20/20, line 9: 20/15, line 10: 20/13, line 11: 20/10.
  the results will be expressed as the mean of the denominator of the Snellen scale (scale 20/--) example. 18.5 ± 1.5, that means the final result is 20/18.5 ± 1.5
Time Frame: 11 days
Population: the analysis by treatment of the research subjects was carried out
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | PRO-156
Number analyzed (Participants) | 30
Number analyzed (eyes) | 60
score on a scale
  basal visit | 19.9 (1.2)
  Final visit | 19.83 (0.9)
Statistical Analysis 1: Comparison: PRO-156; Test type: Other; p = 0.890, Friedman test

2. Secondary Outcome: Intraocular Pressure (IOP)
Description: The tension of a healthy eye should be between 10 and 20 millimeters of mercury (mmHg). In Goldman-type Applying Tonometry, the cornea is flattened, and the intraocular pressure is determined by measuring the force of application and the flattened area.
Time Frame: 11 days
Population: the analysis of the study population was by protocol with Wilcoxon test
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | PRO-156
Number analyzed (Participants) | 30
Number analyzed (eyes) | 60
mmHg
  basal visit | 12.60 (2.47)
  Final visit | 12.23 (2.47)
Statistical Analysis 1: Comparison: PRO-156; Test type: Other; p = 0.078, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Number of Eyes With Epithelial Defects
Description: the number of epithelial defects was evaluated by the application of fluorescein, Staining was performed with fluorescein which stained the degenerated cells and the mucus filaments present in the tear film.
Time Frame: 11 days
Population: the statistical analysis was performed by protocol
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PRO-156
Number analyzed (Participants) | 30
Number analyzed (eyes) | 60
eyes | 0
Statistical Analysis 1: Comparison: PRO-156; Test type: Other; p = 1.000, Friedman test

4. Secondary Outcome: Number of Cases With Adverse Events
Description: The presence of adverse events was evaluated by the number of cases.
Time Frame: 11 days
Population: the statistical analysis was performed by protocol
Measure: Number; unit: cases
Units Other Than Participants: eyes
Arm/Group | PRO-156
Number analyzed (Participants) | 30
Number analyzed (eyes) | 60
cases | 6
Statistical Analysis 1: Comparison: PRO-156; Test type: Other; p = .497, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: The evaluation period was throughout the study (13 days) comprising 11 days of intervention plus 2 days of safety call
Arm/Group | PRO-156
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 6/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO-156 (N=30)
rash (Skin and subcutaneous tissue disorders) | 1 (32) — rash located on the neck and face of the patient of a few hours duration, treated with a single dose of loratadine 10 mg
ocular burning (Eye disorders) | 4 (4)
Tearing (Eye disorders) | 2 (2)
Red Eye (Eye disorders) | 2 (2)
eye pruritus (Eye disorders) | 4 (4)
Foreign body sensation in the eyes (Eye disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
by contract only the sponsor has the rights to the results of the study, if the principal researcher wishes the publication or discuss for dissemination of the same can only perform them prior written authorization with the sponsor and its legal department.